CLINICAL TRIAL: NCT00002306
Title: Multi-Center Evaluation of Fluconazole (UK-49,858) as Treatment for Acute Cryptococcal Meningitis in Patients Who Have Failed to Respond or Have Experienced Unacceptable Toxicity During Treatment With Amphotericin B
Brief Title: A Study of Fluconazole in the Treatment of Cryptococcal Meningitis in Patients Who Have Not Had Success With Amphotericin B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 012I; 056-161
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-02

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Fluconazole; Acquired Immunodeficiency Syndrome; Amphotericin B
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
To evaluate the safety and effectiveness of fluconazole as treatment for acute cryptococcal meningitis in patients who have had an unsatisfactory response to or have experienced unacceptable toxicity with amphotericin B.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Immunosuppressant therapy.
* Antiviral therapy such as zidovudine.
* Prophylaxis for Pneumocystis carinii pneumonia.
* Aerosolized pentamidine.

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Not previously treated for acute cryptococcal meningitis and not eligible for Pfizer Central Research, protocol #159.

* Patients must have a baseline cerebrospinal fluid (CSF) culture-positive for Cryptococcus neoformans.
* Written informed consent must be obtained for each patient, either from the patient himself or from the patient's legal guardian.
* Each individual patient must be approved by Pfizer Central Research prior to study entry.

Prior Medication:

Allowed:

* Immunosuppressant therapy.
* Antiviral therapy such as zidovudine.
* Prophylaxis for Pneumocystis carinii pneumonia.
* Aerosolized pentamidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy to or intolerance of imidazoles or azoles.
* Moderate or severe liver disease.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy to or intolerance of imidazoles or azoles.
* Moderate or severe liver disease.
* Satisfactory response to amphotericin B and have received a total amphotericin B dose of 15 mg/kg or more since CSF culture documentation of the current episode of acute cryptococcal meningitis.
* Life expectancy of < 2 weeks.

Prior Medication:

Excluded:

* Coumadin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.

Prior Treatment:

Excluded:

* Lymphocyte replacement.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of South Florida, Tampa, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - Univ Hosp, Boston, Massachusetts
  - Ann Arbor Veterans Administration Med Ctr, Ann Arbor, Michigan
  - Washington Univ School of Medicine, St Louis, Missouri
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Cincinnati Veterans Adm Med Ctr / Univ Hosp, Cincinnati, Ohio
  - United States Air Force Med Ctr, Lackland Air Force Base, Texas
  - Southwest Texas Methodist Hosp, San Antonio, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas